CLINICAL TRIAL: NCT02546739
Title: Phase I Study of T Cells Expressing an Anti-CD19 Chimeric Receptor in Children and Young Adults With B Cell Malignancies
Brief Title: Immunotherapy With CD19 CAR T-cells for B-Cell Lymphoma, ALL and CLL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Doing Biomedical Co., Ltd. (Industry)
Collaborators: The First Hospital of Jilin University (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doing-002
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; CAR T
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: 1 (Experimental): Acute lymphoblastic leukemia treated with chimeric antigen receptor modified T cells(Anti-CD19-CAR) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR
- Experimental: 2 (Experimental): Chronic lymphoblastic leukemia with chimeric antigen receptor modified T cells(Anti-CD19-CAR) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR
- Experimental: 3 (Experimental): Non-hodgkin lymphoma treated with chimeric antigen receptor modified T cells(Anti-CD19-CAR) targeting CD19.
  Interventions: Biological: Anti-CD19-CAR

INTERVENTIONS:
Biological: Anti-CD19-CAR — Cells extracted, followed by induction chemotherapy before CD19-CAR infusion (dose escalation.)

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of CD19 Chimeric Antigen Receptor (CAR) redirected autologous T-cells in patients with high risk, relapsed CD19+ haematological malignancies.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19 Chimeric Antigen Receptor (CAR) T-cells (CD19 CAR T-cells) in patients with high risk, relapsed CD19+ haematological malignancies (Leukemia and lymphoma). Following informed consent and registration to the trial, patients will undergo an unstimulated leukapheresis for the generation of the CD19 CAR T-cells. Patients will receive the CD19CAR T-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CAR T-cells in patients with high risk relapsed CD19+ malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell derived acute lymphoblastic leukemia(ALL), chronic lymphoblastic leukemia(CLL) and non-hodgkin lymphoma.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 70 years.
5. CD19 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 30% by flow cytometry.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.
12. Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to trial.

Exclusion Criteria:

1. KPS<50.
2. Patients are allergic to cytokines.
3. Central nervous system leukemia within 28 days.
4. Uncontrolled active infection.
5. Acute or chronic GVHD.
6. Treated with T cell inhibitor.
7. Pregnancy and nursing females.
8. HIV/HBV/HCV Infection.
9. Other situations we think improper for the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of each patient. | 3 years
  Determine the toxicity profile of the CD19 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-CD19 CAR T cells in vivo. | 3 years
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Antitumor Effects | Every 3 months post treatment up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.
Maximum tolerated dose (MTD) of CD19 targeted CAR T cells. | 4 weeks
  Maximum tolerated dose (MTD) of CD19 targeted CAR T cells.

CONTACTS AND LOCATIONS:
Overall Officials: li gangyi, master, Study Chair — Beijing Doing Biomedical Co., Ltd.
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hebei Yanda Ludaopei Hospital, Sanhe, Hebei
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huai'An First People'S Hospital, Huaian, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Shanxi Dayi Hospital, Taiyuan, Shanxi
  - Tianjin people's hospital, Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - Beijing DOING Biomedical Co., Ltd, Beijing